CLINICAL TRIAL: NCT07145463
Title: A Prospective, Multicenter, Randomized Controlled Clinical Study Evaluating the VitaFlow Liberty® Flex Transcatheter Aortic Valve Retrievable and Steerable Delivery System for the Treatment of Severe Aortic Stenosis
Brief Title: Prospective, Multicenter, Randomized Controlled Clinical Study Evaluating the VitaFlow Liberty® Flex Transcatheter Aortic Valve Delivery System for the Treatment of Severe Aortic Stenosis Lesions
Acronym: Flex-TAVR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: First Hospital of China Medical University (Other); The Affiliated Hospital of Qingdao University (Other); First Affiliated Hospital of Fujian Medical University (Other); Renmin Hospital of Wuhan University (Other); The First Affiliated Hospital of Nanchang University (Other); The Second Affiliated Hospital of Dalian Medical University (Other); Guangdong Provincial People's Hospital (Other); General Hospital of Ningxia Medical University (Other); Sichuan Provincial People's Hospital (Other); Second Affiliated Hospital of Nanchang University (Other); Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Flex-TAVR trial
Record Dates: First submitted 2025-07-30; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Aortic Valve Stenosis
Keywords: TAVR; Steerable Delivery System; Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Intervention Model Description: This is a prospective, multicenter, randomized controlled study;Randomization will be performed at a 1:1 ratio using a central randomization system;All subjects will undergo clinical follow-up before discharge, at 30 days, and at 1 year post-procedure;An independent data management and statistical center, along with a clinical monitoring organization, will collect, organize, and statistically analyze all relevant clinical data;
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational Device (Experimental): Transcatheter Aortic Valve Retrievable and Controllable Flex Delivery System (VitaFlow Liberty® Flex)
  Interventions: Device: Transcatheter Aortic Valve Replacement
- Control Device (Active Comparator): Transcatheter Aortic Valve and Delivery System (Self-Expanding Valve, Non-Controllable Flex Delivery System)
  Interventions: Device: Transcatheter Aortic Valve Replacement

INTERVENTIONS:
Device: Transcatheter Aortic Valve Replacement — Transcatheter Aortic Valve Implantation/Replacement (TAVI/TAVR) has gradually emerged as a new treatment option for patients with severe aortic stenosis who are ineligible for open-heart valve replacement or at high surgical risk.

SUMMARY:
This is a prospective, multicenter, randomized controlled clinical study designed to evaluate the real-world performance of the VitaFlow Liberty® Flex Transcatheter Aortic Valve Retrievable and Steerable Delivery System (Investigational Device) for treating severe aortic stenosis (AS) in challenging anatomies. The study will compare it against the VitaFlow Liberty® Retrievable Delivery System (Control Device), which lacks steerability.

Key Study Elements:

Objective: The primary objective is to assess the device's performance using the incidence of a composite endpoint before hospital discharge. This endpoint includes permanent pacemaker implantation (PPI), valve-in-valve (ViV) implantation, or moderate-to-severe paravalvular leakage (PVL).

Design: A prospective, multicenter RCT with 1:1 randomization (Experimental: VitaFlow Liberty® Flex vs. Control: VitaFlow Liberty®). Approximately 15 sites in China will participate. Subjects undergo follow-up at discharge, 30 days, and 1 year post-procedure. An independent data center handles management and analysis.

Population: Patients with severe AS (echo confirmed: peak velocity ≥4.0 m/s, mean gradient ≥40 mmHg, or AVA ≤1.0 cm²/AVAi ≤0.6 cm²/m²) AND preoperative CTA showing a challenging aortic-left ventricular angle >60°. NYHA class ≥II is required.

Devices:

Investigational: VitaFlow Liberty® Flex (Retrievable & Steerable Delivery System - Models DSRS21/24/27/30/A series; Loading Tools LT-S series).

Control: VitaFlow Liberty® (Retrievable Delivery System - Models DSR21/24/27/30; Loading Tools LT series).

Endpoints:

Primary: Composite of PPI, ViV, or moderate-to-severe PVL before discharge.

Secondary: Include individual components of the primary endpoint (ViV, PVL) immediately post-procedure, procedural success (VARC-3), technical assistance rates, valve retrievals, implantation depth, arch/valve crossing performance, valve hemodynamics (gradient, area, leak, LVEF), NYHA class, Major Adverse Cardiac and Cerebrovascular Events (MACCE - all-cause death, MI, stroke, reoperation), major vascular complications (at discharge/30 days).

Key Inclusion: Severe AS, challenging anatomy (aortic-LV angle >60°), NYHA ≥II, informed consent.

Key Exclusions: Device/contrast allergies, anticoagulant intolerance, active infection, severe vascular disease prohibiting access, ascending aorta ≥55mm, unsuitable aortic root anatomy, intracardiac mass/thrombus, recent MI (<30 days), severe concomitant mitral/tricuspid regurgitation, cardiogenic shock, severe LV dysfunction (LVEF<20%), hematologic abnormalities, pregnancy/breastfeeding, participation in other device trials.

Visits: Screening (≤30d pre-op), Procedure (intra-op to 24h post-op), Discharge (≤7d post-op), 30d Follow-up (±7d), 12m Telephone FU (±1m).

Sample Size: Planned enrollment of 232 subjects (116 per group), calculated for superiority testing. Based on an expected composite endpoint rate of 21% for the Flex system vs. a historical rate of 38% for non-steerable systems (Superiority margin Δ1=0%, one-sided α=2.5%, Power=80%, accounting for 5% dropout).

Purpose: This study aims to demonstrate the superiority of the retrievable and steerable VitaFlow Liberty® Flex delivery system in reducing the composite rate of key adverse events (PPI, ViV, significant PVL) at discharge compared to the non-steerable system, specifically in patients with severe AS and anatomically challenging aortic-left ventricular angles.

DETAILED DESCRIPTION:
A Prospective, Multicenter, Randomized Controlled Clinical Trial Evaluating the VitaFlow Liberty® Flex Transcatheter Aortic Valve Retrievable and Steerable Delivery System for Severe Aortic Stenosis in Challenging Anatomies

1. Study Rationale and Objective Severe aortic stenosis (AS) carries significant morbidity and mortality when untreated. Transcatheter aortic valve replacement (TAVR) has emerged as a standard therapy, yet complex aortic anatomies - particularly steep aortic-left ventricular (LV) angles - present technical challenges during valve delivery, potentially leading to suboptimal deployment, paravalvular leak (PVL), conduction disturbances requiring permanent pacemaker implantation (PPI), or valve-in-valve (ViV) placement. The VitaFlow Liberty® Flex Delivery System addresses this with its retrievable and steerable catheter technology designed for enhanced navigability. This prospective, multicenter, randomized controlled trial (RCT) aims to evaluate the real-world superiority of the investigational VitaFlow Liberty® Flex System versus the non-steerable VitaFlow Liberty® System in patients with severe AS and challenging anatomies (aortic-LV angle >60°). The primary objective is to compare the incidence of a composite safety endpoint (PPI, ViV implantation, or moderate-to-severe PVL) before hospital discharge.
2. Study Design

Type: Prospective, multicenter, open-label, 1:1 randomized controlled superiority trial

Randomization: Centralized electronic system

Blinding: Unblinded (procedural nature precludes blinding)

Study Arms:

Experimental: VitaFlow Liberty® Flex TAVR System (Retrievable & Steerable)

Control: VitaFlow Liberty® TAVR System (Retrievable, Non-Steerable)

Follow-up Schedule:

Pre-discharge (≤7 days post-op)

30 days (±7 days)

12 months (±1 month, telephone)

Oversight: Independent Clinical Events Committee (CEC), Data Monitoring Committee (DMC), and Core Laboratories for imaging/ECG analysis

Centers: ~15 experienced TAVR centers across China

3. Investigational and Control Devices

Device Component：VitaFlow Liberty® FLEX (Investigational) VitaFlow Liberty® (Control) Delivery System Type：Retrievable & Steerable(Investigational) Retrievable (Non-Steerable)(Control)

4. Study Population

Diagnosis: Severe symptomatic AS confirmed by echocardiography:

Peak aortic velocity ≥4.0 m/s OR Mean gradient ≥40 mmHg OR Aortic valve area (AVA) ≤1.0 cm² (or AVAi ≤0.6 cm²/m²) Anatomical Inclusion: Pre-op CT angiography (CTA) with 3D reconstruction demonstrating aortic-LV angle >60° (validating challenging anatomy).

Symptoms: NYHA Functional Class ≥II.

Key Exclusion Criteria:

Allergy to device materials (nitinol), contrast, or antiplatelets/anticoagulants Active infection/endocarditis Severe vascular disease prohibiting access Ascending aorta diameter ≥55mm Unsuitable aortic root anatomy (e.g., heavy calcification affecting expansion) Intracardiac thrombus/mass Recent MI (<30 days) Severe mitral/tricuspid regurgitation LVEF <20% Hematologic disorders (leukopenia, thrombocytopenia, coagulopathy) Pregnancy or concurrent device trials

5. Endpoints

Primary Endpoint:

Composite of PPI, ViV implantation, or moderate-to-severe PVL before discharge.

Secondary Endpoints:

Procedural:

ViV rate (immediate post-op) Moderate-to-severe PVL (immediate post-op) Technical assistance crossing rate Valve retrieval attempts Valve implantation depth Arch/valve crossing performance Procedural success (VARC-3 criteria*)

Clinical:

PPI rate (discharge, 30 days) MACCE** (discharge, 30 days): All-cause death, MI, stroke, reoperation Major vascular complications

Hemodynamic/Echocardiographic:

Valve orifice area, mean gradient, peak velocity Degree of stenosis/regurgitation LVEF (immediate, discharge, 30 days)

Functional: NYHA Class improvement (discharge, 30 days)

*VARC-3: Valve Academic Research Consortium-3 criteria for technical success.

**MACCE: Major Adverse Cardiac and Cerebrovascular Events.

6. Statistical Analysis & Sample Size Hypothesis: Superiority of VitaFlow Liberty® Flex

Assumptions:

Historical composite endpoint rate (non-steerable systems): 38% Expected composite rate (steerable system): 21% Superiority margin (Δ1): 0% Power: 80% | One-sided α: 2.5% | Dropout: 5% Sample Size: 232 subjects (116 per arm)

Analysis:

Primary endpoint: Chi-square/Fisher's exact test Secondary endpoints: Mixed-effects models accounting for site variability Subgroup analyses: Valve size, center volume, baseline aortic-LV angle

7. Study Procedures

Screening (≤30 days pre-op): Echocardiography, CTA, NYHA assessment, informed consent.

Procedure: TAVR under standard anesthesia. Randomization pre-insertion. Discharge (≤7 days): Echo, ECG, NYHA, MACCE/vascular complication assessment. 30-Day Visit: Clinical exam, echo, ECG, lab tests, NYHA, MACCE. 12-Month Follow-up: Telephone assessment for mortality/MACCE.

8. Ethical & Regulatory Considerations

Approved by institutional review boards (IRBs) at all sites. Conducted per ICH-GCP, Declaration of Helsinki, and Chinese regulatory requirements.

Independent DMC reviews safety data quarterly.

9. Significance and Innovation

This trial addresses a critical unmet need in TAVR: improving outcomes in patients with challenging aortic anatomies. If superiority is demonstrated, the steerable delivery system may become the preferred option for:

Reducing PPI rates (linked to anatomical precision) Mitigating PVL (via optimal deployment) Avoiding ViV (through recapture/repositioning) Enhancing first-attempt success in tortuous anatomies

Conclusion:

This rigorously designed RCT will provide Level A evidence on the clinical utility of steerable TAVR technology in high-risk anatomies, potentially establishing a new standard for managing complex AS patients.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of severe aortic stenosis, defined as: echocardiographically confirmed peak aortic valve velocity ≥4.0 m/s, or mean aortic valve gradient ≥40 mmHg, or aortic valve area (AVA) ≤1.0 cm2 (or AVA index ≤0.6 cm2/m2);
2. Preoperative cardiac and great vessel CT angiography (CTA) with 3D reconstruction demonstrating an aortic-left ventricular angle >60°, indicating potential challenges for arch crossing and valve crossing;
3. New York Heart Association (NYHA) functional class ≥II;
4. Voluntary participation in the study with signed informed consent.

Exclusion Criteria:

1. Known allergy or intolerance to components of the investigational or control devices (e.g., nitinol) or contrast agents;
2. Contraindication or known allergy to anticoagulant or antiplatelet therapy, rendering the patient unable to tolerate such treatment;
3. Known active infective endocarditis or other active infections;
4. Known severe vascular disease that would preclude safe prosthetic valve implantation;
5. Ascending aorta width ≥55mm;
6. Pre-procedural imaging shows aortic root anatomy unsuitable for transcatheter aortic valve implantation (including aortic root calcification that may affect proper valve expansion);
7. Pre-procedural echocardiography shows intracardiac mass, left ventricular or left atrial thrombus, or vegetation;
8. Acute myocardial infarction within 30 days prior to procedure (defined as Q-wave MI or non-Q-wave MI);
9. Concomitant severe mitral or tricuspid regurgitation;
10. Concomitant cardiogenic shock or hemodynamic instability requiring inotropic support, mechanical ventilation, or mechanical cardiac assistance;
11. Concomitant severe left ventricular dysfunction (defined as left ventricular ejection fraction LVEF<20%);
12. Concomitant hematologic abnormalities defined as leukopenia (WBC count <3×109/L), thrombocytopenia (platelet count <30×109/L), history of bleeding diathesis or coagulopathy, or hypercoagulable state;
13. Female subjects known to be pregnant or breastfeeding;
14. Subjects currently participating in or planning to participate in other drug or device clinical studies within 12 months postoperatively; Any other condition that the investigator or heart team deems may hinder the subject's safe participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
the number of occurrences/total number of occurrences | Perioperative/Periprocedural"
  Incidence of composite endpoint events before discharge (permanent pacemaker implantation, valve-in-valve, or moderate-to-severe paravalvular leak) calculated as number of occurrences/total number of occurrences

SECONDARY OUTCOMES:
Incidence of valve-in-valve | Perioperative/Periprocedural
  Incidence of valve-in-valve calculated as: Occurred/Total
Incidence of Moderate-to-severe paravalvular leak | Perioperative/Periprocedural
  Incidence of Moderate-to-severe paravalvular leak calculated as: Occurred/Total
Incidence of Other technical assistance crossing rate | Perioperative/Periprocedural
  Incidence of Other technical assistance crossing rate (immediately post-procedure) calculated as: Occurred/Total
Incidence of valve retrievals | Perioperative/Periprocedural
  Incidence of valve retrievals calculated as: Occurred/Total
Valve implantation depth calculated as Intraoperative images | Perioperative/Periprocedural
  Valve implantation depth calculated as Intraoperative images
Incidence of Permanent Pacemaker Implantation | Perioperative/Periprocedural, 30 days,
  Incidence of Permanent Pacemaker Implantation calculated as: Occurred/Total
Arch Crossing and Valve Crossing Performance calculated as assessment scale | Perioperative/Periprocedural
  Arch Crossing and Valve Crossing Performance calculated as assessment scale
Number of participants with Valve Performance Evaluation | Perioperative/Periprocedural, 30 days,
  Valve Performance Evaluation, Including: Valve Orifice Area, Mean Transvalvular Pressure Gradient, Peak Transvalvular Velocity, Degree of Valve Stenosis, Degree of Valve Regurgitation, Degree of Paravalvular Leak, Left Ventricular Ejection Fraction (LVEF) calculated as cardiac uhrasonography
NYHA Functional Class Assessment NYHA classification | Perioperative/Periprocedural, 30 days
  NYHA Functional Class Assessment NYHA classification: Divided into four levels, Grade I: No discomfort in daily activities, and no restriction in physical activities. Grade II: Mild activity restriction, no symptoms at rest, but daily activities (such as climbing stairs) can cause fatigue and palpitation. Grade III: obvious activity limitation, no symptoms at rest, but slight activity (such as walking) will cause symptoms. Grade Ⅳ: There are symptoms at rest, and any activity aggravates discomfort.
Incidence of Major Adverse Cardiac and Cerebrovascular Events (MACCE) | Perioperative/Periprocedural, 30 days,
  Incidence of Major Adverse Cardiac and Cerebrovascular Events (MACCE)，MACCE Includes: All-Cause Mortality, Myocardial Infarction, All Stroke, Reoperation Due to Valve Dysfunction calculated as: Occurred/Total
Incidence of Major Vascular Complications | Perioperative/Periprocedural, 30 days
  Incidence of Major Vascular Complications calculated as: Occurred/Total
Procedural Success Rate (VARC-3 Definition) | Perioperative/Periprocedural
  Procedural Success Rate (VARC-3 Definition) calculated as: Occurred/Total

CONTACTS AND LOCATIONS:
Overall Officials: Wenzhi Pan, MD, Study Chair — Fudan University
Locations (1):
- 180 Fenglin Road, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Cribier A, Eltchaninoff H, Bash A, Borenstein N, Tron C, Bauer F, Derumeaux G, Anselme F, Laborde F, Leon MB. Percutaneous transcatheter implantation of an aortic valve prosthesis for calcific aortic stenosis: first human case description. Circulation. 2002 Dec 10;106(24):3006-8. doi: 10.1161/01.cir.0000047200.36165.b8. PMID 12473543
- [Background] Grube E, Laborde JC, Gerckens U, Felderhoff T, Sauren B, Buellesfeld L, Mueller R, Menichelli M, Schmidt T, Zickmann B, Iversen S, Stone GW. Percutaneous implantation of the CoreValve self-expanding valve prosthesis in high-risk patients with aortic valve disease: the Siegburg first-in-man study. Circulation. 2006 Oct 10;114(15):1616-24. doi: 10.1161/CIRCULATIONAHA.106.639450. Epub 2006 Oct 2. PMID 17015786
- [Result] Supino PG, Borer JS, Preibisz J, Bornstein A. The epidemiology of valvular heart disease: a growing public health problem. Heart Fail Clin. 2006 Oct;2(4):379-93. doi: 10.1016/j.hfc.2006.09.010. No abstract available. PMID 17448426
- [Result] Carabello BA, Paulus WJ. Aortic stenosis. Lancet. 2009 Mar 14;373(9667):956-66. doi: 10.1016/S0140-6736(09)60211-7. Epub 2009 Feb 21. PMID 19232707
- [Result] Leon MB, Smith CR, Mack M, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Brown DL, Block PC, Guyton RA, Pichard AD, Bavaria JE, Herrmann HC, Douglas PS, Petersen JL, Akin JJ, Anderson WN, Wang D, Pocock S; PARTNER Trial Investigators. Transcatheter aortic-valve implantation for aortic stenosis in patients who cannot undergo surgery. N Engl J Med. 2010 Oct 21;363(17):1597-607. doi: 10.1056/NEJMoa1008232. Epub 2010 Sep 22. PMID 20961243